CLINICAL TRIAL: NCT00002329
Title: A Randomized, Placebo-Controlled, Double-Blind, Single and Multiple Oral Dose-Tolerance Study of Oral MDL 28,574A Solution in HIV-Positive Patients
Brief Title: A Study of MDL 28,574A in HIV-Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoechst Marion Roussel (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 221A; NDPR0002
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1995-05

CONDITIONS: HIV Infections
Keywords: MDL 28574
MeSH Terms: conditions — HIV Infections | interventions — celgosivir

INTERVENTIONS:
Drug: Celgosivir hydrochloride

SUMMARY:
To characterize the safety profile of MDL 28574A following both acute and subchronic dosing in HIV-positive patients. To determine the MTD of both acute and subchronic doses of this drug when administered as oral solution. To determine the pharmacokinetic profile of MDL 28574A and castanospermine (from which MDL 28574A is derived) following both acute and subchronic dosing.

DETAILED DESCRIPTION:
In Part A of the study, patients receive a single oral dose of MDL 28574A on day 1 and are followed through day 7. In Part B, patients receive single daily doses of the drug on days 1 through 14 and are followed through day 21.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection.
* CD4 count >= 500 cells/mm3.
* No evidence of AIDS.
* No antiretroviral therapy within 30 days prior to study entry.

NOTE:

* Presence of lymphadenopathy in two or more extrainguinal sites, at least 1 cm in diameter for 3 or more months, is permitted.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Clinically significant abnormalities on routine hematology (other than CD4 count and Western blot), serum chemistry, and urinalysis.
* Abnormal EKG.
* Positive stool guaiac.
* Abnormal medical history or physical exam including temperature, heart rate, and blood pressure.
* Clinically significant organ abnormality or disease.
* Positive urine drug screen for illicit drugs.
* Inability to comply with study procedures.

Concurrent Medication:

Excluded:

* Routine treatment with nonprescription medications.
* Treatment with other medications except with approval of the investigator.

Patients with the following prior conditions are excluded:

* Prior participation in this trial.
* Serious physical or mental illness within 1 year prior to study entry that would confound interpretation of data.

Prior Medication:

Excluded:

* Antiretroviral therapy within 30 days prior to study entry.
* Known medications that alter renal, hepatic, or hematologic/immunologic function (such as barbiturates, phenothiazines, cimetidine, and immunomodulators) within 14 days prior to study entry.
* Routine treatment with nonprescription medications within 3 days prior to study entry.

History of alcohol or drug abuse within the past year.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Francis Mem Hosp, San Francisco, California, United States